CLINICAL TRIAL: NCT03641131
Title: A Retrospective, Post-Marketing, Sentinel-based Active Surveillance Study to Evaluate the Safety of Ampholipad Using Real-World Data in Taiwan
Brief Title: Ampholipad Real-World Data in Taiwan
Status: Completed | Type: Observational
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Other Study IDs: TLC166B4013
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Aspergillus Infection; Febrile Neutropenia; Candida Infection; Fungal Infection; Cryptococcal Infections
MeSH Terms: conditions — Aspergillosis; Febrile Neutropenia; Candidiasis; Mycoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective, post-marketing, multi-center chart review study includes patients who had been prescribed Ampholipad.

DETAILED DESCRIPTION:
A retrospective, post-marketing, multi-center chart review study includes patients who had been prescribed Ampholipad in selected sentinel hospitals in Taiwan. Medical charts of approximately 100 treated patients will be reviewed by the investigators to collect the pre-specified data, including indication, underlying cancer type (only for cancer patients), demographics, and concomitant medications as well as all the laboratory examination data regarding renal function from 1 month prior to first dose of Ampholipad up to 1 week after the last dose of the initial treatment course.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 2 years of age
2. Patients who had received at least one dose of Ampholipad treatment, with available baseline serum creatinine (SCr) data within 1 month prior to first Ampholipad use and at least one post baseline SCr data during treatment period

Exclusion Criteria:

1. Patients whose medical chart cannot provide both the start and stop dates of Ampholipad for a course of treatment (first course only)
2. Patients who had documented HIV infection diagnosis
3. Patients with potential end-stage renal disease (ESRD) receiving regular dialysis within 1 month prior to first Ampholipad use

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had received at least one dose of Ampholipad treatment in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Incidence of nephrotoxicity | Ampholipad treatment course, up to 42 days
  Nephrotoxicity is defined as an increase in serum creatinine (SCr) to >2X baseline value and the post-baseline peak SCr > 1.2 mg/dL

SECONDARY OUTCOMES:
Proportion of SCr >1.5X, SCr >2X or SCr >3X of the baseline values | From 1 month prior to first dose of Ampholipad up to 1 week after the last dose of the initial treatment course
  Incidence of SCr >1.5X, SCr >2X or SCr >3X of the baseline values
Incidence of Adverse Drug Reaction (ADR) | From 1 month prior to first dose of Ampholipad up to 1 week after the last dose of the initial treatment course
  Number of ADRs reported/collected during the protocol-defined retrospective medical chart review period
eGFR | From 1 month prior to first dose of Ampholipad up to 1 week after the last dose of the initial treatment course
  Changes in estimated glomerular filtration rate (eGFR) from baseline throughout the Ampholipad treatment period
Survival rate | From 1 month prior to first dose of Ampholipad up to 1 week after the last dose of the initial treatment course
  Survival rate through 7 days after the last day of the Ampholipad treatment
Microbiological eradication rate | From 1 month prior to first dose of Ampholipad up to 1 week after the last dose of the initial treatment course
  Microbiological eradication rate of Ampholipad treatment
Fever resolution rate | From 1 month prior to first dose of Ampholipad up to 1 week after the last dose of the initial treatment course
  Fever resolution rate of Ampholipad treatment in febrile neutropenic patients

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, PhD, Study Director — Taiwan Liposome Company
Locations (6):
- Taiwan (6):
  - Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Hospital, Tainan
  - Taipei Municipal Wanfang Hospital, Taipei
  - Tri Service General Hospital, Taipei

REFERENCES:
- [Background] Girois SB, Chapuis F, Decullier E, Revol BG. Adverse effects of antifungal therapies in invasive fungal infections: review and meta-analysis. Eur J Clin Microbiol Infect Dis. 2005 Feb;24(2):119-30. doi: 10.1007/s10096-005-1281-2. PMID 15711785
- [Background] Laniado-Laborin R, Cabrales-Vargas MN. Amphotericin B: side effects and toxicity. Rev Iberoam Micol. 2009 Dec 31;26(4):223-7. doi: 10.1016/j.riam.2009.06.003. PMID 19836985
- [Background] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of America. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2011 Feb 15;52(4):e56-93. doi: 10.1093/cid/cir073. PMID 21258094
- [Background] White MH, Bowden RA, Sandler ES, Graham ML, Noskin GA, Wingard JR, Goldman M, van Burik JA, McCabe A, Lin JS, Gurwith M, Miller CB. Randomized, double-blind clinical trial of amphotericin B colloidal dispersion vs. amphotericin B in the empirical treatment of fever and neutropenia. Clin Infect Dis. 1998 Aug;27(2):296-302. doi: 10.1086/514672. PMID 9709879
- [Background] Wingard JR, White MH, Anaissie E, Raffalli J, Goodman J, Arrieta A; L Amph/ABLC Collaborative Study Group. A randomized, double-blind comparative trial evaluating the safety of liposomal amphotericin B versus amphotericin B lipid complex in the empirical treatment of febrile neutropenia. L Amph/ABLC Collaborative Study Group. Clin Infect Dis. 2000 Nov;31(5):1155-63. doi: 10.1086/317451. Epub 2000 Nov 7. PMID 11073745
- [Background] Walsh TJ, Finberg RW, Arndt C, Hiemenz J, Schwartz C, Bodensteiner D, Pappas P, Seibel N, Greenberg RN, Dummer S, Schuster M, Holcenberg JS. Liposomal amphotericin B for empirical therapy in patients with persistent fever and neutropenia. National Institute of Allergy and Infectious Diseases Mycoses Study Group. N Engl J Med. 1999 Mar 11;340(10):764-71. doi: 10.1056/NEJM199903113401004. PMID 10072411